CLINICAL TRIAL: NCT05945199
Title: Effectiveness of tDCS on Reducing Craving in Patients Practicing Chemsex: a Single-center, Double-blind, Randomized Controlled Pilot Trial
Acronym: CHEMSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PETIT AOI 2021
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Chemsex
MeSH Terms: conditions — Chemsex | interventions — Transcranial Direct Current Stimulation; Weights and Measures

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS active (Experimental)
  Interventions: Device: tDCS; Behavioral: Assessment of risk behaviours; Other: Scales
- Sham tDCS (Placebo Comparator)
  Interventions: Device: tDCS; Behavioral: Assessment of risk behaviours; Other: Scales

INTERVENTIONS:
Device: tDCS — * 1 session/day for 5 consecutive days
  * stimulation at an intensity of 2 mA for the active tDCS group and sham stimulation (using the device's sham mode) for the placebo group
Behavioral: Assessment of risk behaviours — Assessment of risk behaviours (retrospective exploration by the categorical rating of frequency: At least once a day - Several times a week several times a week - once a week - several times a month - once a month - less than once a month - never). times a month - Once a month - Less than once a month - Never)
Other: Scales — EVA craving index for chemsex Maximum VAS craving in the week preceding assessment for chemsex, sexual practices and use of psychoactive substances, HAqII, CSBD-19, modified CCQ-brief, SDI, BDI-II

SUMMARY:
The aim of this research is to evaluate the efficacy of a new treatment for chemsex or "chemical sex", the use of psychoactive substances to modify sexual experience and performance. This treatment, called Transcranial direct current stimulation (tDCS) aims to modulate the cortical activity of brain areas involved in the desire to use psychoactive substances, or drugs, and the desire for uncontrolled sexual intercourse.

This treatment should therefore lead to a reduction in the craving for consumption of psychoactive substances and/or the practice of uncontrolled sexual activity.

The stakes of this new treatment are high, because chemsex exposes people to health risks for themselves and others. These risks include the risk of infection (skin infections, HIV infection, hepatitis viruses), psychological harms (anxiety attacks, depression, suicide risk), risk of addiction (addiction to the psychoactive product used, sex addiction), and toxicological harm (overdose, dangerous combination of psychoactive substances) or trauma (blows, trauma to the genitals or anorectal trauma).

To date, there is no proven therapeutic treatment for people wishing to reduce or stop chemsex.

40 participants will be randomized into 2 groups:

* 20 patients will receive active stimulation
* 20 patients will receive sham stimulation

The total duration of the study for each patient will be 13 weeks: 1 week of stimulation and 12 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient who provides written consent
* Patient aged ≥ 18 years
* Patient motivated and willing to change chemsex behavior, assessed by examiner during screening and inclusion visits
* Patient using at least one of the following psychoactive substances to modify sexual performance and/or experience:

  * Cathinones, or methamphetamine, or MDMA, or cocaine, or ketamine, or GBL/GHB
  * ≥ 1 time per month over the past 6 months and/or ≥ 10 times over the past year

Exclusion Criteria:

* Patient with a substance use disorder not involved in the practice of chemsex
* Patient with a recent change (< 1 month) in the prescription of a psychotropic treatment
* Patient presenting an acute psychiatric condition requiring hospitalization and/or immediate modification of a psychotropic treatment
* Patients with unstable or uncontrolled neuropsychiatric disease
* Patients with a history of epileptic seizures
* Patients with unexplained episodes of loss of consciousness, as this condition may be linked to cerebral alterations or epilepsy
* Patients with advanced or decompensated somatic pathology, requiring hospitalization expected during study follow-up
* Patients suffering from any serious life-threatening illness, such as congestive heart failure, chronic obstructive pulmonary disease or active neoplasia
* Patients with implanted cerebral medical devices, implanted pacemakers, or any electrically, magnetically or mechanically activated implant.
* Patients with cardiac, neural or drug implants
* Patients with vascular clips or other electrically sensitive support systems in the brain
* Patients with severe brain lesions
* Patients with skin lesions at stimulation sites
* Patients with skin problems such as dermatitis, psoriasis or eczema
* Patients with severe or frequent headaches
* Patients who have already benefited from tDCS sessions
* Pregnant, parturient or breast-feeding women (pregnancy test)
* Staff working in the addictology department of Dijon University Hospital
* Patient participating in another clinical trial
* Patient not affiliated to national health insurance
* Patient unable to complete assessment scales
* Patient under psychiatric care without consent or under legal protection (guardianship, curatorship)
* Major incapable or unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Assessment of cue-induced craving for chemsex using a visual analogue scale | 4 weeks from end of stimulation (S5)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France